CLINICAL TRIAL: NCT05186168
Title: The Corin MiniHip and Trinity Advanced Bearing Acetabular Cup System UK Clinical Surveillance Study
Brief Title: Corin MiniHip and Trinity Cup Clinical Surveillance Study
Status: Active, not recruiting | Type: Observational
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: MH101
Record Dates: First submitted 2021-12-15; First posted 2022-01-11 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Total Hip Arthroplasty; Osteoarthritis, Hip; Traumatic Arthritis of Hip; Rheumatoid Arthritis of Hip; Developmental Dysplasia of the Hip; Avascular Necrosis of the Femoral Head
MeSH Terms: conditions — Osteoarthritis, Hip; Developmental Dysplasia of the Hip; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MiniHip Stem — The MiniHip stem is a titanium femoral stem (Ti-6Al-4V) coated with a layer of hydroxyapatite applied over a layer of pure titanium
Device: Trinity Acetabular Cup System — The Trinity Acetabular System is a modular acetabular cup system consisting of a press fit, titanium alloy shell

SUMMARY:
The aim of the study is to provide long term follow up data on the performance and safety of the Corin MiniHip and Trinity acetabular cup over a 10-year period.

DETAILED DESCRIPTION:
To verify the ten-year clinical and radiographic performance of the Corin MiniHip and Trinity Advanced Bearing Acetabular System when used in patients under normal conditions of use.

To document the safety, evaluate patient satisfaction, quality of life and to determine the survivorship following intervention with the Corin MiniHip and Trinity Advanced Bearing Acetabular System at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* A severely painful and/or disabled joint from osteoarthritis, traumatic arthritis, rheumatoid arthritis or developmental dysplasia of the hip.
* Avascular necrosis of the femoral head
* All subjects must be between the age of 18 and 75 at the time of surgery to take part in this study
* Scheduled for a primary total hip replacement.

Exclusion Criteria:

* Active infection
* Severe Obesity (BMI over 35)
* Pregnancy
* Mental illness
* Grossly distorted anatomy (surgeon's discretion)
* Sepsis
* Osteomyelitis
* Osteomalacia
* Distant foci of infections
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Muscular atrophy or neuromuscular disease
* Allergy to implant material
* Marked bone loss or bone resorption
* Patients without sufficient quantities of synovial fluid to allow for proper lubrication, such as patients with Sjogren's syndrome
* Skeletally immature patients and cases where there is a loss of abductor musculature, poor bone stock or poor skin coverage around the hip joint which would make the procedure inappropriate
* Any case not described in the inclusion criteria
* Any patient who cannot or will not provide informed consent for participation in the study
* Those whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suitable participants undergoing primary total hip replacement with the Corin MiniHip and Trinity Advanced Bearing Acetabular System.
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2011-03-15 (Actual); Primary Completion 2028-05-03 (Estimated); Study Completion 2028-05-03 (Estimated)

PRIMARY OUTCOMES:
Post operative survivorship of the Minihip Stem and Trinity acetabular Cup system at 10-year follow-up | 10 years
  Survivorship measured via Kaplan-Meier (KM) curve

SECONDARY OUTCOMES:
Harris Hip Score (HHS) up to 10-year follow-up | Baseline to 10 years
  Harris Hip Score is a disease-specific scoring system, originally intended as an outcome score after arthroplasty surgeries that includes the domains of function, pain, motion and deformity. Minimum score is 0, Maximum score is 100. The score is reported as 90-100 for excellent results, 80-89 for good, 70-79 for fair, 60-69 for poor, and below 60 for a failed result.
Oxford Hip Score (OHS) up to 10-year follow-up | Baseline to 10 years
  Oxford Hip Score is a patient-centered questionnaire that is designed to assess functional ability and pain from the patient's perspective. It is a short, twelve-item questionnaire developed for completion by patients undergoing THA. Minimum score 0 indicating worst outcome, maximum score 48 indicating best outcome.
Hip- and device-related adverse events up to 10-year follow-up | Baseline to 10 years
  All hip-related and device-related complications, including those occurring during the surgical procedure and throughout the postoperative evaluations, are required to be documented and reviewed
Trinity acetabular cup radiographic performance up to 10-years | Baseline to 10 years
  Radiographic assessment considering Acetabular radiolucent lines using the De lee Charney measurement of zones 1 - 3.
Minihip Stem radiographic performance up to 10-years | Baseline to 10 years
  Radiographic assessment considering osteolysis and femoral stem alignment measured as Varus/Valgus and the use of the Gruen's assessment zones 1-7
Minihip Stem and Trinity acetabular cup radiographic performance up to 10-years | Baseline to 10 years
  Radiographic assessment considering heterotopic ossifications using the Brooker classification Grade 1 - 4.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Field, Principal Investigator — Elective Orthopaedic Centre, Epsom Hospital, Epsom, Surrey, KT18 7EG